CLINICAL TRIAL: NCT07067047
Title: The Effect of Nursing Care Decision Support System Designed for Fluid Volume Excess of Patients With Heart Failure on Clinical Outcomes of Patients and Home Self-Care Outcomes
Acronym: HF-DSS-Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leyla Biçen (Other)
Responsible Party: Sponsor-Investigator, Leyla Biçen, PhD Candidate in Public Health Nursing, Ege University, Institute of Health Sciences, Ege University
Organization: Ege University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0219; NotApplicable (Other: Not Applicable - The study was not funded by any agency.)
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing Decision Support System Group (Experimental)
  Interventions: Behavioral: Nursing Decision Support System

INTERVENTIONS:
Behavioral: Nursing Decision Support System — A behavioral intervention involving a nurse-led decision support system designed to manage fluid volume overload in heart failure patients. The intervention guided nursing care planning, monitoring, and evaluation during hospitalization and through home follow-up visits.

SUMMARY:
This study aims to evaluate the effects of a nursing care decision support system designed to reduce fluid overload in patients with heart failure. The goal is to examine its impact on clinical outcomes both during hospitalization and after discharge at home. The study focuses on improving nursing interventions and patient follow-up through structured, evidence-based decision-making tools.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heart failure (HF)
* Aged 18 years or older
* Ejection fraction below 50%
* Presence of +1 or greater pitting edema in the extremities
* Voluntary agreement to participate in the study
* Sufficient cognitive and communicative ability to participate in interviews and complete scales/forms

Exclusion Criteria:

* Presence of additional comorbidities other than cardiac risk factors (e.g., dialysis-dependent renal failure, lymphedema, oncology patients, etc.)
* Presence of severe valvular stenosis
* History of amputation
* Classified as morbidly obese
* Isolated right heart failure
* Inadequate cooperation or communication skills
* Terminal stage patients
* Absence of echocardiographic evaluation
* BNP level not measured

Criteria for Discontinuation During the Study:

* Inaccessible by phone
* Withdrawal of consent
* Development of poor general condition during follow-up
* Transferred to intensive care units during follow-up
* Extended hospitalization due to infection or other secondary causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Congestion Score Improvement | Baseline to 30 days post-discharge
  Assessment of the reduction in fluid volume overload symptoms based on a standardized congestion scoring system. The score evaluates parameters such as edema, shortness of breath, and weight changes.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University Atatürk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No